CLINICAL TRIAL: NCT03298685
Title: SAFETIM Besoins: Suivi Des Adolescents Des Familles et Des Equipes Pour Une Transition Idéale en Mucoviscidose Etude Des Besoins Adolescents et Parent Avant après Transition
Brief Title: SAFETIM-needs : Exploring Adolescent's and Parent's Needs During Transition in French CF Centers
Acronym: SAFETIM-needs
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.005; 2017-A00062-51 (Other: ID RCB)
Record Dates: First submitted 2017-08-01; First posted 2017-10-02 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis; Adolescent Behavior
Keywords: transition; care program; needs
MeSH Terms: conditions — Cystic Fibrosis; Adolescent Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patient and parents cohort in 3 CF center: All adolescents for whom the transition to the adult center is scheduled within six months and their parent will be interviewed before and after transition.
  Interventions: Other: semi structured interviews for all adolescents and their parent

INTERVENTIONS:
Other: semi structured interviews for all adolescents and their parent — Before and after transition, individual semi structured interviews will be recorded by one person in the same way in all CF center. And every interview will be transcribed by an other person

SUMMARY:
prospective multicentric study protocol in french CF center, exploring adolescent avec parents needs during transition from pediatric CF center to adult CF center

DETAILED DESCRIPTION:
Adolescent's and parent's needs will be studied, before the transition and their experiences of transition, in order to propose organizational national recommendations semi structured interview with adolescents and parents separately, before and after transition.

semi structured interviews will be conducted twice for each (adolescent and parents), the first in the 6 months before transition and the second in the 6 months after transition.

After their verbatims will be analyzed and the optimal organisation will be determined for the transition based according to their point of view.

At the end, the data from this study will be matched with data collected in a former study from care givers practices during transition in the french CF centers.

ELIGIBILITY:
Inclusion Criteria:

* CF adolescent and their parents , for whom the transition to the adult center is scheduled within six months and witch have freely agreed to participate in the interviews

Exclusion Criteria:

* none

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: CF adolescent and their parents , for whom the transition to the adult center is scheduled within six months and witch have freely agreed to participate in the interviews their age will be between 17 and 23 years old. living followed in one of the 3 CF center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Identify CF adolescents and their parents needs before transition | During their systematic appointment at the CF center, patients will have one individual interview during the year before transition. Interviews will be analyzed after all interviews will have been performed.
  Qualitative analysis of interviews
Identify CF adolescents and their parents experience after transition | During their systematic appointment at the CF center, patients will have one individual interview during the year after transition. Interviews will be analyzed after all interviews will have been performed.
  Qualitative analysis of interviews

SECONDARY OUTCOMES:
What do they need, to feel safe before transition | During their systematic appointment at the CF center, patients and parents will have one individual interview during the year before transition. Interviews will be analyzed after all interviews will have been performed
  Identify patients and parents needs
Do these needs of CFadolescent and their parents taken into account in the transition procedures | During their systematic appointment at the CF center, patients and parents will have one individual interview during the year after transition. Interviews will be analyzed after all interviews will have been performed
  Do the procedures take into account the needs of patients and parents
Which factors influence quality of transition other than TPE dimension. | Interviews will be analyzed after an average of one year after the last interviews will have been performed, both outcome will be matched
  Satisfaction level of Patients and Family After Transition
Do the resources implemented by the CRCM teams during the adolescent-adult transition matched with adolescents and parents needs and expectations | comparison between the results with health care practices one year after the last interview will be performed
  Identifying key points of the patient's personalized transition, the timing and personalization of the health care course during the transition

CONTACTS AND LOCATIONS:
Overall Officials: LLERENA catherine, MD, Principal Investigator — CHU GA Grenobe France
Locations (4):
- France (4):
  - University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - UniversityHospitalGrenoble, Grenoble
  - Hôpital Femme Mère Enfant, HCL, Lyon
  - South Hospital of Lyon, HCL, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bregnballe V, Schiotz PO, Lomborg K. Parenting adolescents with cystic fibrosis: the adolescents' and young adults' perspectives. Patient Prefer Adherence. 2011;5:563-70. doi: 10.2147/PPA.S25870. Epub 2011 Nov 7. PMID 22114471
- [Background] Kreindler JL, Miller VA. Cystic fibrosis: addressing the transition from pediatric to adult-oriented health care. Patient Prefer Adherence. 2013 Dec 11;7:1221-6. doi: 10.2147/PPA.S37710. PMID 24376344
- [Background] Blum RW, Garell D, Hodgman CH, Jorissen TW, Okinow NA, Orr DP, Slap GB. Transition from child-centered to adult health-care systems for adolescents with chronic conditions. A position paper of the Society for Adolescent Medicine. J Adolesc Health. 1993 Nov;14(7):570-6. doi: 10.1016/1054-139x(93)90143-d. No abstract available. PMID 8312295
- [Background] Sawicki GS, Lukens-Bull K, Yin X, Demars N, Huang IC, Livingood W, Reiss J, Wood D. Measuring the transition readiness of youth with special healthcare needs: validation of the TRAQ--Transition Readiness Assessment Questionnaire. J Pediatr Psychol. 2011 Mar;36(2):160-71. doi: 10.1093/jpepsy/jsp128. Epub 2009 Dec 29. PMID 20040605
- [Background] Davis AM, Brown RF, Taylor JL, Epstein RA, McPheeters ML. Transition care for children with special health care needs. Pediatrics. 2014 Nov;134(5):900-8. doi: 10.1542/peds.2014-1909. Epub 2014 Oct 6. PMID 25287460